CLINICAL TRIAL: NCT06622382
Title: Bariatric Endoscopic Antral Myotomy (BEAM) for Weight Loss - a Pilot Study
Brief Title: BEAM for Weight Loss - a Pilot Study
Acronym: BEAM pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stephen KK Ng, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2024.223
Record Dates: First submitted 2024-09-21; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bariatric endoscopic antral myotomy (Experimental): Bariatric endoscopic antral myotomy (BEAM) is a novel endoscopic technique which is performed using a gastroscope under general anesthesia. It involves cutting the muscle fibers at the gastric antrum, thereby weakening the antral pump, delaying gastric emptying and inducing satiety.
  Interventions: Procedure: Bariatric endoscopic antral myotomy

INTERVENTIONS:
Procedure: Bariatric endoscopic antral myotomy — A mucosal incision is performed using a triangle-tip knife J at the level of the incisura along the level of the greater curvature. Submucosal tunneling is then performed and stopped immediately proximal to the pylorus. Two parallel lines of partial thickness myotomy are then performed from the distal to proximal antrum using the same endoscopic knife. The myotomy is stopped approximately 2 cm distal to the mucosal incision site. Finally, the mucosal incision is closed using endoclips after haemostasis is confirmed.

SUMMARY:
Bariatric endoscopic antral myotomy (BEAM) is a novel endoscopic technique which is performed using a gastroscope under general anesthesia. It involves cutting the muscle fibers at the gastric antrum, thereby weakening the antral pump, delaying gastric emptying and inducing satiety. Early reports had shown that this technique can produce significant weight loss. Furthermore, this technique has the potential benefits of lower risks, improved durability and allows subsequent mucosal assessment of stomach, which is important in Asia countries with higher prevalence of gastric intestinal metaplasia or gastric cancers. Given that this novel endoscopic technique has not been widely adopted for treatment of obesity, this pilot study aims to investigate the efficacy and safety of BEAM in obese patients who are eligible for endoscopic bariatric therapies.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal or more than 30kg/m2 (27.5kg/m2 for Chinese or South Asian) to 40kg/m2, or BMI equal or more than 40kg/m2 and patient is either high risk for surgery or unwilling to undergo surgery, AND
* failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone or in combination

Exclusion Criteria:

* Previous upper GI surgery (e.g. bariatric surgery, anti-reflux surgery; gastrectomy; esophageal surgery)
* Gastroparesis
* Active smoking
* An ongoing or a history of treatment with opioids in the last 12 months prior to enrollment
* Previous pyloromyotomy or pyloroplasty
* Gastrointestinal obstruction
* Use of any medication that may interfere with weight loss or gastric emptying
* Severe coagulopathy
* Esophageal or gastric varices and/or portal hypertensive gastropathy
* Underlying uncontrolled endocrine problem that leads to obesity. (e.g. Hypothyroidism, Cushing syndrome, eating disorder etc.)
* Any inflammatory disease of the gastrointestinal tract (including but not limited to severe (LA Grade C or D) esophagitis, active gastric ulceration, active duodenal ulceration, or specific inflammation such as Crohn's disease)
* Malignancy
* Pregnant or breast feeding
* Patients not fit for general anesthesia
* ASA grade IV or V
* Mental or psychiatric disorder; Drug or alcohol addiction
* Other cases deemed by the examining physician as unsuitable for safe treatment
* Refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | baseline, 1,3,6,12 months
  Weight change compared to baseline
Adverse events | within 30 days of procedure
  Adverse events relating to endoscopic intervention, graded according to the Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Technical success rate | 1 day
  successful completion of endoscopic procedures
Serum ghrelin levels | baseline, 1,3,6,12 months
  Serum ghrelin levels compared to baseline
Blood pressure | baseline, 1,3,6,12 months
  Blood pressure and anti-hypertensive medication use compared to baseline
Lipid profile | baseline, 1,3,6,12 months
  Lipid profile compared to baseline
Pain scale after procedure | 3 days
  measured by visual analogue scale (0:no pain - 10:worst pain)
Change in Quality of Life | baseline, 1,6,12 months
  measured by 36-Item Short Form Survey (SF-36) questionnaire - (0:worst - 100:best)
Gastric emptying symptoms | baseline, 1,6,12 months
  measured by gastroparesis cardinal symptom index (GCSI) - (0:best - 45:worst)
Fasting glucose level | baseline, 1,3,6,12 months
  levels compared to baseline
Insulin level | baseline, 1,3,6,12 months
  levels compared to baseline
HbA1c level | baseline, 1,3,6,12 months
  levels compared to baseline
serum liver parameters | baseline, 1,3,6,12 months
  AST, ALT, ALP and GGT level compared to baseline
hepatic steatosis index | baseline, 1,3,6,12 months
  level compared to baseline
NAFLD fibrosis | baseline, 1,3,6,12 months
  NAFLD fibrosis scores compared to baseline (F0: no liver fibrosis - F4: significant liver fibrosis)
obstructive sleep apnea | baseline, 1,3,6,12 months
  Change in sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ng, FRCSEd(Gen), Principal Investigator — Prince of Wales Hospital, the Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided